CLINICAL TRIAL: NCT00373581
Title: Effects of Vigabatrin on Cocaine Self-Administration
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding ran out
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Novel Cocaine Pharmacotherapies (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5096; DA 10755 (Other Grant/Funding Number: Novel Cocaine Pharmacotherapies)
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Cocaine Dependence
Keywords: Vigabatrin; GABA levels; Smoked cocaine
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Vigabatrin; Cocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vigabatrin, cocaine (Experimental)
  Interventions: Drug: Vigabatrin; Drug: Cocaine
- placebo, cocaine (Placebo Comparator)
  Interventions: Drug: Vigabatrin; Drug: Cocaine

INTERVENTIONS:
Drug: Vigabatrin
Drug: Cocaine

SUMMARY:
The objective of this study is to determine if vigabatrin will decrease cocaine self-administration, cardiovascular effects, subjective effects and craving compared to placebo.

DETAILED DESCRIPTION:
Two recent open label clinical trials have reported that the anticonvulsant, gamma vinyl-GABA (GVG; vigabatrin), decreases relapse to cocaine use (Brodie et al., 2003, 2005). Vigabatrin increases neural GABA levels by irreversibly inhibiting the primary GABA degradation enzyme, GABA-transaminase; the hypothesized mechanism by which vigabatrin decreases cocaine relapse is by increasing GABA levels, thereby decreasing the effects of cocaine and cocaine-associated environmental cues on extracellular dopamine concentrations in the mesolimbic dopaminergic pathway (Morgan and Dewey, 1998). We are proposing to use our model of repeated dose cocaine self-administration to assess the interaction between vigabatrin and smoked cocaine under controlled laboratory conditions. This 57-day outpatient/inpatient /outpatient/inpatient protocol will evaluate the effects of vigabatrin maintenance (0, 3 g/day) on cocaine craving, subjective effects, and self-administration using a within-subjects design. Non-treatment seeking cocaine-dependent volunteers will be maintained outpatient for 14 days of vigabatrin maintenance prior to beginning each inpatient study phase. During the inpatient phases, volunteers will live on a hospital clinical research unit and will participate in laboratory sessions in which they will have the opportunity to purchase doses of smoked cocaine (0, 12, 25, 50 mg; $5/administration). In addition to measuring cocaine self-administration, we will measure the cardiovascular and subjective effects of repeated cocaine administration and cocaine craving under each vigabatrin maintenance condition. Determining vigabatrin's effects on a range of smoked cocaine doses will provide essential data on the mechanism of the vigabatrin-cocaine interaction.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for current cocaine abuse
* Average use of smoked cocaine is at least 2x/week for past 6 mos; currently spends at least $70 per week on cocaine
* Has patterns of smoked cocaine use in terms of frequency and amounts which parallel or exceed those administered in the study
* Age 21-45
* Able to give informed consent, and comply with study procedures
* Agrees to practice an effective form of contraception

Exclusion Criteria:

* Current seizure disorder or heart disease
* Currently meeting DSM-IV criteria for all major psychiatric/psychotic disorders. Volunteers with a history of depression or psychosis will also be excluded (p. 43, Investigator's brochure)
* Dependence on substances other than cocaine or nicotine
* Request for drug treatment
* Judged to be noncompliant with study protocol
* Clinical laboratory tests outside normal limits that are unacceptable to the study physician (e.g., BP > 140/90; BUN, creatinine, LFTs > 1.5 ULN; hematocrit < 34 for women, < 36 for men; pseudocholinesterase deficiency)
* Current parole or probation
* Recent history of significant violent or suicidal behavior
* Pregnancy or lactation
* Baseline visual field defects

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2006-04; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Subjective effects
Cardiovascular effects
Cravings
Cocaine Administration

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Haney, Ph.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- Irving Center for Clinical Research, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No